CLINICAL TRIAL: NCT02221596
Title: Vitamin D Contribution to Muscle Metabolic Function in Aged Adults
Brief Title: Vitamin D and Muscle Metabolic Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Travis Thomas (Other)
Responsible Party: Sponsor-Investigator, David Travis Thomas, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: 1R21AG046762-01A1 (NIH)
Record Dates: First submitted 2014-08-14; First posted 2014-08-20 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: Vitamin D; 25(OH)D; Aerobic training; Near-infrared spectroscopy; Diffuse correlation spectroscopy; MRS
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- vitamin D + aerobic training (Experimental): vitamin D capsules every weekday (10,000IU/day) and exercise
  Interventions: Dietary Supplement: vitamin D; Other: aerobic training
- vitamin D + no aerobic training (Active Comparator): vitamin D capsules every weekday (10,000IU/day) and no exercise
  Interventions: Dietary Supplement: vitamin D
- placebo + aerobic training (Active Comparator): placebo capsule every weekday and exercise
  Interventions: Other: aerobic training
- placebo + no aerobic training (No Intervention): placebo capsule every weekday and no exercise

INTERVENTIONS:
Dietary Supplement: vitamin D — 50,000IU/wk of vitamin D3
  Arms: vitamin D + aerobic training; vitamin D + no aerobic training
Other: aerobic training — 7 days of treadmill training during the 13th week of study
  Arms: placebo + aerobic training; vitamin D + aerobic training

SUMMARY:
The purpose of this study is to identify the magnitude of muscle lipid redistribution and muscle oxygen use in individuals 60 years old or older following combined treatment of vitamin D repletion and aerobic training compared to vitamin D repletion alone, aerobic training alone, or no treatment.

DETAILED DESCRIPTION:
The investigators plan to recruit approximately 56 aged individuals with vitamin D insufficiency for a 13 week trial. All subjects will be 60 years of age or older. Participants will be randomized to one of four groups: vitamin D (50,000IU/wk) + aerobic training (7 days during the 13th week); vitamin D (50,000IU/wk) + normal daily activity during the 13th week; placebo + aerobic training (7 days during the 13th week); or placebo + normal daily activity during the 13th week.

Following screening and informed consent process a physical activity questionnaire will be administered. A blood draw will then be conducted at baseline, midpoint and endpoint. Collected blood for the purposes of this study will assess vitamin D status (25(OH)D), parathyroid hormone, ionized calcium, insulin, and a comprehensive metabolic panel. At baseline and endpoint muscle lipid will be assessed using Magnetic Resonance Spectroscopy and muscle oxygen consumption will be determined using a novel hybrid diffuse optical instrument consisting of a near-infrared spectroscopy and a diffuse correlation spectroscopy. In addition, at each study time point 3 dietary recalls will be completed and physical activity will be measured using an accelerometer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60 and older
* BMI: 18.5-29
* Communicates fluently in English

Exclusion Criteria:

* Metal implant not suitable for MRI
* Any form of hormone replacement therapy
* Engage in more than 1 hr/week of vigorous activity
* Participated in a high-intensity resistance or aerobic training program in the last 3 months
* Lower extremity injury or surgery in the past 3 months
* Foot sores or bone conditions severely limiting ability to move or perform exercise or joint pain made worse by mild exercise
* Diabetes, inflammatory bowel disease, renal disease or uncontrolled hypertension.
* Currently have or had a history of cardiovascular or pulmonary disease that would preclude the involvement in the performance of exercise
* History of myopathy (including congenital myopathies)
* History of neurological conditions related to spinal derangement, disk disease, peripheral neuropathies, tremor and rigidity
* Past medical history of hyperparathyroidism, kidney stones or rhabdomyolysis
* Currently receiving treatment for vitamin D deficiency
* Vitamin D level >30ng/mL
* Currently smoking

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
blood measure | Change from Baseline in vitamin D at 13 weeks
  vitamin D

SECONDARY OUTCOMES:
muscle lipid | baseline and 13 weeks after baseline
  Intramyocellular lipid and extramyocellular lipid will be assessed using magnetic resonance spectroscopy and fat segmentation.
muscle oxygen consumption | baseline and 13 weeks after baseline
  Local muscle tissue oxidative capacity will be measured using a novel hybrid diffuse optical instrument consisting of a near-infrared spectroscopy (NIRS) and a diffuse correlation spectroscopy (DCS)

CONTACTS AND LOCATIONS:
Overall Officials: D. Travis Thomas, Ph.D., RD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States